CLINICAL TRIAL: NCT01855984
Title: Tocotrienols Supplementation in School Going Children With Attention Deficit/Hyperactivity Disorder(ADHD) - A Randomized Controlled Trial
Brief Title: Tocotrienols for School-going Children With ADHD
Acronym: TOCAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RCSI & UCD Malaysia Campus (Other)
Collaborators: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, May Loong Tan, Dr, RCSI & UCD Malaysia Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRR-6767
Record Dates: First submitted 2013-05-10; First posted 2013-05-17 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Children; Tocotrienol
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral mixed tocotrienols (Experimental): 2 capsules containing 100mg mixed tocotrienols per capsule taken orally once a day for 6 months
  Interventions: Dietary Supplement: Oral mixed tocotrienols
- Placebo (Placebo Comparator): 2 capsules containing soya bean oil taken orally once a day for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral mixed tocotrienols — 200mg per day
  Other Names: Tocovid Suprabio.
  Arms: Oral mixed tocotrienols
Dietary Supplement: Placebo — Capsules containing soya bean oil that has similar appearance with the mixed tocotrienol capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if tocotrienol supplementation given to school going children with ADHD will result in reduction of their ADHD symptoms.

DETAILED DESCRIPTION:
The main objective of the study is to:

a. Determine if supplementation of tocotrienol compared to placebo has an effect on the symptoms of school going children with ADHD.

The secondary objective is to:

1. Determine if supplementation of tocotrienol compared to placebo has an effect on the dose of current medication used in school going children with ADHD.
2. Determine the safety of tocotrienol in the study population.
3. Determine if tocotrienol levels in children with ADHD correlate with their symptom scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD in accordance with the Diagnostic and Statistical Manual (DSM) IV criteria.
* Be able to swallow soft gel capsules.
* If already on medication for ADHD, the dose of the medication must be stable for the last 3months
* Be able to attend all follow up visits.
* Be agreeable to have their teacher score the National Initiative for Children's Healthcare Quality (NICHQ) Vanderbilt Assessment Scale - Teacher Informant
* Be willing to have their blood taken 3 times during the study.

Exclusion Criteria:

* ADHD caused by syndromes, inborn errors of metabolism, or structural brain lesions.
* Co-existing chronic liver disease
* Current use of anticoagulant or antiplatelet drugs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ADHD symptom scores as measured by NICHQ Vanderbilt Parent and Teacher Assessment Scales | Change of total symptom scores from baseline at 6 months

SECONDARY OUTCOMES:
Change in the dose of current medication for ADHD | After 6 months intervention
Number of participants with adverse reaction | 6 months
Blood tocotrienol levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: May Loong Tan, MRCPCH(UK), Principal Investigator — RCSI & UCD Malaysia Campus
Locations (1):
- Child & Adolescent Psychiatry Unit, Hospital Pulau Pinang, George Town, Pulau Pinang, Malaysia